CLINICAL TRIAL: NCT01577199
Title: Randomized Prospective Controlled Non-inferiority Trial of Low-dose Clomiphene Based Antagonist Protocol vs. High Dose Gonadotropin/Antagonist Protocol for IVF Poor Responders
Brief Title: RCT of Low-dose Clomiphene vs. High Dose Gonadotropin Protocol for IVF Poor Responders
Acronym: CLOVANT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: no subjects recruited
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1112012095
Record Dates: First submitted 2012-04-11; First posted 2012-04-13 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Infertility
Keywords: IVF; poor responder; low ovarian reserve; ART; ovarian stimulation; IVF protocols
MeSH Terms: conditions — Infertility | interventions — Clomiphene; Gonadotropins; follitropin alfa; follitropin beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High dose gonadotropins (Active Comparator): High dose gonadotropins protocol compared to Low-dose Clomiphene
  Interventions: Drug: High dose gonadotropins
- Low-dose Clomiphene (Experimental): clomid-based, low dose gonadotropin protocol compared to High dose gonadotropins
  Interventions: Drug: Low-dose Clomiphene

INTERVENTIONS:
Drug: Low-dose Clomiphene — Pretreatment with a 0.1mg estradiol patch in the luteal phase starting 10 days after the LH surge followed by clomiphene citrate 100mgon days 2-6 of the menstrual cycle with 225 international units of gonadotropins (eg Follistim , Menopur) starting on day 5
  Other Names: clomiphene citrate with low dose gonadotropins
  Arms: Low-dose Clomiphene
Drug: High dose gonadotropins — Pretreatment with a 0.1mg estradiol patch in the luteal phase starting 10 days after the LH surge followed high dose gonadotropins (eg. Follistim. Menopur) 600IU starting on day 2 of the cycle
  Other Names: Gonal F or Follistim
  Arms: High dose gonadotropins

SUMMARY:
The purpose of this study is compare two commonly-used medication protocols ( low-dose clomiphene citrate and high dose gonadotropin protocols) for the treatment of patients with diminished ovarian reserve (decreased number of eggs remaining in the ovary) undergoing IVF. This research is being done because we do not know if these two medication protocols are equally likely to help a woman become pregnant.

DETAILED DESCRIPTION:
The objective of this protocol is to prospectively evaluate whether a clomid-based, low dose gonadotropin protocol (225 IU) would be non-inferior in terms of mature oocyte yield (eggs that are ready to be fertilized) as compared to a high-dose protocol.

Patients meeting the criteria for poor ovarian response will be consented and randomized to either a stimulation protocol involving pretreatment with a 0.1mg estradiol patch in the luteal phase starting 10 days after the LH surge (the hormone released by the brain to cause ovulation to occur, which is detectable in urine) followed by oral clomiphene citrate 100mg on days 2-6 of the menstrual cycle and 225 international units of gonadotropins starting on day 5, or to the control group involving the same pretreatment with 0.1mg luteal estradiol patches starting 10 days after the LH surge, with high dose gonadotropins (600IU) alone, starting on day 2 of the cycle. After randomization, patients will undergo routine IVF procedures, monitoring, blood draws, cancellation criteria, oocyte retrieval, and embryo transfer as non-study participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18-42 undergoing IVF
* AFC <7 (see definition above) and AMH (see definition above) <0.5 and/or prior poor IVF response

Exclusion Criteria:

* BMI (body mass index) >30
* PGD (preimplantation genetic diagnosis, in which embryos are biopsied to rule out chromosomal abnormalities)
* Age >42
* Fragile X carriers (a condition associated with premature ovarian aging)
* TESE (Testicular sperm extraction)
* Asherman's syndrome (uterine scarring which can affect implantation and pregnancy)
* Untreated hydrosalpinx (accumulated fluid in the fallopian tube which may be toxic to embryos)
* >6 prior attempted cycles

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The number of mature oocytes retrieved | 1 year
  To evaluate the number of mature oocytes retrieved in two different IVF protocols for poor responders

SECONDARY OUTCOMES:
The number of embryos transferred | 1year
  To evaluate the number of embryos transferred

CONTACTS AND LOCATIONS:
Overall Officials: Owen Davis, MD, Principal Investigator — WCMC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Center for Reproductive Medicine — http://www.IVF.org